CLINICAL TRIAL: NCT02350569
Title: A Phase 2, Multicenter, Open-Label Study to Investigate the Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed Dose Combination Administered in Patients Infected With Chronic HCV for Use in the Peri-Operative Liver Transplantation Setting
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed Dose Combination Administered in Patients Infected With Chronic Genotype 1 or 4 HCV for Use in the Peri-Operative Liver Transplantation Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1428
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C Virus Infection
Keywords: liver transplant; hepatitis C; Gilead; Communicable Diseases; Infection; Liver Diseases; RNA Virus Infections
MeSH Terms: conditions — Hepatitis C; Communicable Diseases; Infections; Liver Diseases; RNA Virus Infections | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LDV/SOF (Experimental): Participants with genotype 1 or 4 HCV who are undergoing liver transplant will receive one dose of LDV/SOF prior to the transplant and then will receive LDV/SOF once daily for 4 weeks following the transplant.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objective of this study is to evaluate the antiviral efficacy of treatment with ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) therapy at the time of liver transplantation and through 4 weeks posttransplant in adults with genotype 1 or 4 hepatitis C virus (HCV) infection who are undergoing primary liver transplantation.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent or for those individuals where hepatic encephalopathy affects their ability to provide initial or ongoing consent, has an appropriate and legally-authorized representative (LAR) willing and able to provide consent on behalf of the individual.
* HCV RNA infection with quantifiable virus at screening
* Must have chronic genotype 1 or 4 HCV infection for ≥ 6 months by medical history or liver biopsy
* Currently on the liver transplantation wait list
* Screening electrocardiogram (ECG) without clinically significant abnormalities.
* A negative serum pregnancy test result is required for females

Key Exclusion Criteria:

* Any previous solid organ transplant
* Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with participant's treatment, assessment, or compliance
* HIV infection or a positive hepatitis B virus surface antigen result
* History of malignancy (with exception of hepatocellular carcinoma within Milan criteria, certain resolved skin cancers or other early cancer for which surgical resection is considered to be completely curative)
* Treatment with any approved or experimental medication with known anti-HCV activity within 1 month prior to screening date
* Prior exposure to an HCV non-structural protein (NS)5A inhibitor
* Patients on hemodialysis prior to or at the time of transplantation will be excluded
* Creatinine clearance (CLcr) < 40 mL/min at screening or < 40 mL/min on day of transplant
* Participation in a clinical study with an investigational drug or biologic within 28 days prior to screening visit
* Receipt or planned receipt of an organ from an HCV positive donor

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2016-03-28 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - San Francisco, California
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Detroit, Michigan
  - New York, New York
  - Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Levitsky J, Verna EC, O'Leary JG, Bzowej NH, Moonka DK, Hyland RH, Arterburn S, Dvory-Sobol H, Brainard DM, McHutchison JG, Terrault NA. Perioperative Ledipasvir-Sofosbuvir for HCV in Liver-Transplant Recipients. N Engl J Med. 2016 Nov 24;375(21):2106-2108. doi: 10.1056/NEJMc1611829. No abstract available. PMID 27959735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 22 May 2015. The last study visit occurred on 22 April 2016.
Pre-assignment Details: 36 participants were screened. 17 unique participants were enrolled into the study (3 received the Day -1 dose and had their transplant cancelled; 2 of these patients were re-enrolled into the Main Study; the 3rd was rescreened but not transplanted).
Groups:
- LDV/SOF: LDV/SOF for 1 Day: 3 participants were called for transplant, received one dose of ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg), but had their liver transplant cancelled. All 3 participants were rescreened and 2 were subsequently re-enrolled, transplanted, and continued into the Main Study.
  Main Study (LDV/SOF 4 Weeks): One dose of ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) immediately prior to receiving a liver transplant, followed by LDV/SOF (90/400 mg) once daily for 4 weeks following transplant in participants with chronic genotype 1 hepatitis C virus (HCV) infection.
  Retreatment (LDV/SOF 12 Weeks): Participants who completed treatment in the Main Study and experienced virologic failure had the option to be retreated with LDV/SOF for 12 weeks.
Period: Main Study (LDV/SOF 4 Weeks)
Arm/Group | LDV/SOF
Started | 16
Completed | 16 (1 participant discontinued treatment, but completed follow-up visits and study.)
Not Completed | 0
Period: Retreatment (LDV/SOF 12 Weeks)
Arm/Group | LDV/SOF
Started | 1 (1 completed treatment (Main Study), experienced virologic failure, and entered Retreatment Phase)
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug during the Main Study
Groups:
- Main Study (LDV/SOF 4 Weeks): One dose of LDV/SOF (90/400 mg) immediately prior to receiving a liver transplant, followed by LDV/SOF (90/400 mg) once daily for 4 weeks following transplant in participants with chronic genotype 1 HCV infection
Arm/Group | Main Study (LDV/SOF 4 Weeks)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 11
  Genotype 1b | 5
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 5
    CT | 9
    TT | 2
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.6 (0.75)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 10
  ≥ 800,000 IU/mL | 6
Prior HCV Treatment [Count of Participants; unit: Participants]
  No | 9
  Yes | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled into the study, received a liver transplant while on study, and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study (LDV/SOF 4 Weeks)
Number analyzed (Participants) | 16
percentage of participants | 87.5 [61.7 to 98.4]

2. Primary Outcome: Percentage of Participants Who Prematurely Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 4 weeks
Population: Safety Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Main Study (LDV/SOF 4 Weeks)
Number analyzed (Participants) | 16
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With SVR 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study (LDV/SOF 4 Weeks)
Number analyzed (Participants) | 16
percentage of participants | 87.5 [61.7 to 98.4]

4. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * End of treatment virologic failure:
    * Completed 28 days LDV/SOF treatment and had HCV RNA ≥ LLOQ at last measurement on treatment
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment HCV RNA measurement.
Time Frame: Up to Posttreatment Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Main Study (LDV/SOF 4 Weeks)
Number analyzed (Participants) | 16
percentage of participants | 6.3

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ While on Treatment at Days 1, 3, 5, 7, 14, 21, and 28
Time Frame: Days 1, 3, 5, 7, 14, 21, and 28
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study (LDV/SOF 4 Weeks)
Number analyzed (Participants) | 16
percentage of participants
  Day 1 | 0 [0.0 to 20.6]
  Day 3 | 12.5 [1.6 to 38.3]
  Day 5 | 18.8 [4.0 to 45.6]
  Day 7: number analyzed (Participants) | 15
  Day 7 | 33.3 [11.8 to 61.6]
  Day 14: number analyzed (Participants) | 15
  Day 14 | 93.3 [68.1 to 99.8]
  Day 21: number analyzed (Participants) | 15
  Day 21 | 100.0 [78.2 to 100.0]
  Day 28: number analyzed (Participants) | 15
  Day 28 | 100.0 [78.2 to 100.0]

ADVERSE EVENTS:
Time Frame: LDV/SOF for 1 Day: After pre-dose to minimum of 30 days or restart of LDV/SOF; Main Study: After pretransplant dose up to 4 weeks plus 30 days; Retreatment: After pretransplant dose up to 12 weeks plus 30 days
Description: Safety Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Groups:
- LDV/SOF for 1 Day: Adverse events reported in this group include participants who received LDV/SOF on Day -1, but did not receive a liver transplant. All 3 participants were rescreened, but only 2 were re-enrolled, transplanted, and received LDV/SOF for 4 weeks.
- Main Study (LDV/SOF 4 Weeks): Adverse events reported in this group include participants with chronic genotype 1 HCV infection who received one dose of LDV/SOF (90/400 mg) prior to receiving a liver transplant, followed by LDV/SOF (90/400 mg) once daily for 4 weeks following transplant.
- Retreatment (LDV/SOF 12 Weeks): Adverse events reported in this group include 1 participant who completed treatment and experienced virologic failure in the Main Study and was retreated with an additional 12 weeks of LDV/SOF.
Arm/Group | LDV/SOF for 1 Day | Main Study (LDV/SOF 4 Weeks) | Retreatment (LDV/SOF 12 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/16 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 5/16 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 14/16 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF for 1 Day (N=3) | Main Study (LDV/SOF 4 Weeks) (N=16) | Retreatment (LDV/SOF 12 Weeks) (N=1)
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Incision site cellulitis (Infections and infestations) | 0 | 1 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Hepatic artery flow decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF for 1 Day (N=3) | Main Study (LDV/SOF 4 Weeks) (N=16) | Retreatment (LDV/SOF 12 Weeks) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 5 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 2 | 0
Ocular icterus (Eye disorders) | 0 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1
Constipation (Gastrointestinal disorders) | 0 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 0
Chills (General disorders) | 0 | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 5 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 3 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 7 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 5 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 5 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Micturition frequency decreased (Renal and urinary disorders) | 0 | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 5 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years